CLINICAL TRIAL: NCT04098640
Title: Molecular Profiling Using FoundationOne CDx in Young (<50 Years of Age) Patients With Metastatic Breast Cancer (ML41263)
Brief Title: Molecular Profiling in Young (<50 Years of Age) Patients With Metastatic Breast Cancer
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Seock-Ah Im, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SNUH_FMI
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
Keywords: Young patient; Asian
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FMI (Other): FoundationOne CDx will be performed using archival tumor tissue
  Interventions: Genetic: FoundationOne CDx

INTERVENTIONS:
Genetic: FoundationOne CDx — FoundationOne CDx will be performed using archival tumor tissue

SUMMARY:
Breast cancer is the most common cancer in women worldwide, especially in developed countries. In developing countries, including South Korea, the incidence and mortality rate of breast cancer is rapidly increasing. One of the most important characteristics of breast cancer in South Korea, as well as in other Asian countries, is the younger onset of disease compared to Western.

Medical treatment of breast cancer is evolving rapidly, incorporating immune checkpoint blockades and molecularly targeted agents. However, data and knowledge are still limited in terms of molecular characteristics of Asian breast cancer, compared to that of Western countries, and this remains a major hurdle for drug development in Asian breast cancer patients.

The primary objective of this study is to elucidate the genetic characteristic of young (<50 years of age) Korean patients with metastatic breast cancer using FoundationOne CDx.

DETAILED DESCRIPTION:
Secondary Objective(s):

1. To evaluate the prognostic and predictive role of tumor mutation burden.
2. To reveal the correlation between genetic characteristics and immunohistochemical expression of selected proteins (including DNA damage repair (DDR) molecules and various immune modulating molecules including PD-L1, PD-1, IDO, and OX40).
3. Compare molecular characteristics of breast cancer according to age groups (<35 years vs. 35-50 years).
4. To offer genomic profiling guided therapy to patients as early as possible (preferably, 1st- or 2nd-line of treatment). In addition, to explore how genomic profiling guided therapy could improve patient outcome as an ad-hoc if sufficient number of patients can be followed up (compared to historic data).

ELIGIBILITY:
Inclusion Criteria:

* Patients between 19 - 50 years of age on the day of signing informed consent.
* Able to provide written informed consent for voluntary participation in the trial.
* With metastatic breast cancer
* Willing to provide biopsies from the primary tumor or lymph nodes at screening to the central laboratory. (with at least 10 unstained slides and 1 H&E slide)

Exclusion Criteria:

* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-09-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Genetic characteristic of young (<50 years of age) Korean patients with metastatic breast cancer. | After the end of patient enrollment
  Genetic characteristics will be evaluated using FoundationOne CDx.

SECONDARY OUTCOMES:
Evaluate the prognostic and predictive role of tumor mutation burden | After the end of patient enrollment
  Tumor mutation burden will be analysed using FoundationOne CDx.
Reveal the correlation between genetic characteristics and immunohistochemical expression of selected proteins. | After the end of patient enrollment
  FoundationOne CDx results and immunohistochemical expression will be analysed.
Compare molecular characteristics of breast cancer according to age groups. | After the end of patient enrollment
  Genetic characteristics will be analysed according to age groups.
To offer genomic profiling guided therapy to patients To explore how genomic profiling guided therapy could improve patient outcome as an ad-hoc if sufficient number of patients can be followed up (compared to historic data). | After the end of patient enrollment
  The result of FoundationOne CDx will be used in patient treatment

CONTACTS AND LOCATIONS:
Overall Officials: Seock-Ah Im, MD PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No